CLINICAL TRIAL: NCT03884738
Title: Effects Of Different Strengthening Methods On Hamstring Muscle Group's Passive Mechanical Properties in Healthy Individuals
Brief Title: Strengthening Effect on Hamstring's Passive Mechanical Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgün Uysal, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HacettepeSportsPhysio
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Sports Physical Therapy
Keywords: Muscle Tonus; Elasticity; Electric Stimulation Therapy; Physical Conditioning, Human
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: randomization into three groups and measurement before and after intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concentric (Active Comparator): Leg Curl Training
  Interventions: Other: Concentric Exercise
- Eccentric (Active Comparator): Nordic Hamstring Training
  Interventions: Other: Nordic Eccentric exercise
- Neuromuscular Electrical Stimulation (Active Comparator): Stimulation Training
  Interventions: Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Concentric Exercise — Leg Curl Machine: 1st week - 1st day is 10 maximum repeat test. 2nd week - 2 days of training - 2 sets of 6 repeats. %60 percent of maximum load.
  3rd week - 3 days of training - 3 sets of 6-8 repeats. %60-80 of maximum load. 4th-8th week - 3 days of training - 3 sets of 8-12 repeats. when 3 sets of 12 achieved, load was increased with 2.5kg.
  Arms: Concentric
Other: Nordic Eccentric exercise — 1. st week - 1 day - 2 sets of 5 repeats.
  2. nd week - 2 days - 2 sets of 6 repeats.
  3. rd week - 3 days - 3 sets of 6-8 repeats.
  4. th week - 3 days - 3 sets of 8-10 repeats. 5-8th weeks - 3 days - 3 sets of 12-8 repeats. When achieved 3 sets of 12 repeats with full range, speed was increased.
  Arms: Eccentric
Other: Neuromuscular Electrical Stimulation — 8 weeks, three times per week, 15 minutes of bilateral hamstring stimulation. 100 Hz. frequency, 600 microsecond duration rectangular current
  Arms: Neuromuscular Electrical Stimulation

SUMMARY:
The purpose of this study was to investigate effects of different strengthening methods on hamstring muscle group's passive mechanical properties and to investigate this effect's relation with performance changes in healthy individuals. 42 healthy sedentary male participated in this study. Passive mechanical properties and strength of hamstring and quadriceps muscles, flexibility of hamstring muscles, anaerobic explosive strength, reaction time, agility were measured. Participants randomized evenly into one of three groups; eccentric, concentric and neuromuscular electrical stimulation (NMES). After 8 weeks training period, participants were measured again.

ELIGIBILITY:
Inclusion Criteria:

* being sedentary

Exclusion Criteria:

* Having knee, hip and/or back pain
* Having a cardiovascular condition/disease
* History of previous knee and/or hip surgery
* Having a diagnose of any systemic disease
* History of previous hamstring injury
* Being physically active within last year ( Regular activity at least 3 days a week and continuity of at least 2 months was accepted as being physically active)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only male participants were accepted
Enrollment: 42 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Passive Mechanical Properties | Change from baseline passive mechanical properties at 8 weeks
  Tone, Elasticity and Stiffness evaluation. Evaluated with Myotonometer-3

SECONDARY OUTCOMES:
Flexibility Measurement | Change from baseline flexibility at 8 weeks
  Sit and reach test was used for hamstring flexibility
Muscle Strength Measurement | Change from baseline muscle strength at 8 weeks
  Hamstring and Quadriceps strength were measured with LaFayette Manuel Muscle Tester
Agility Measurement | Change from baseline agility time at 8 weeks
  Illinois Agility Test was used for agility measurement
Anaerobic Explosive Power | Change from baseline anaerobic explosive power at 8 weeks
  Jump and Reach test was administered
Reaction Time | Change from baseline reaction time at 8 weeks
  ruler drop test was used for reaction timing

CONTACTS AND LOCATIONS:
Overall Officials: tuzun fırat, Assoc. Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayala F, Sainz de Baranda P, De Ste Croix M, Santonja F. Reproducibility and criterion-related validity of the sit and reach test and toe touch test for estimating hamstring flexibility in recreationally active young adults. Phys Ther Sport. 2012 Nov;13(4):219-26. doi: 10.1016/j.ptsp.2011.11.001. Epub 2012 Jan 23. PMID 23068896
- [Background] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Background] Amiri-Khorasani M, Sahebozamani M, Tabrizi KG, Yusof AB. Acute effect of different stretching methods on Illinois agility test in soccer players. J Strength Cond Res. 2010 Oct;24(10):2698-704. doi: 10.1519/JSC.0b013e3181bf049c. PMID 20168255
- [Background] Schwesig R, Koke A, Fischer D, Fieseler G, Jungermann P, Delank KS, Hermassi S. Validity and Reliability of the New Handball-Specific Complex Test. J Strength Cond Res. 2016 Feb;30(2):476-86. doi: 10.1519/JSC.0000000000001061. PMID 26815176
- [Background] Mjolsnes R, Arnason A, Osthagen T, Raastad T, Bahr R. A 10-week randomized trial comparing eccentric vs. concentric hamstring strength training in well-trained soccer players. Scand J Med Sci Sports. 2004 Oct;14(5):311-7. doi: 10.1046/j.1600-0838.2003.367.x. PMID 15387805
- [Background] Glaviano NR, Langston WT, Hart JM, Saliba S. Influence of patterned electrical neuromuscular stimulation on quadriceps activation in individuals with knee joint injury. Int J Sports Phys Ther. 2014 Dec;9(7):915-23. PMID 25540707